CLINICAL TRIAL: NCT05009953
Title: An Open-label, Multicentre, Phase II Study to Evaluate the Safety and Efficacy of Irinotecan Liposome Injection in Patients With Advanced Biliary Tract Cancer
Brief Title: Study of Irinotecan Liposome Injection in Patients With Advanced Biliary Tract Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Internal strategy change. Not related to safety concerns.
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE072-CSP-003
Record Dates: First submitted 2021-08-04; First posted 2021-08-18 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Advanced Biliary Tract Cancer; Intrahepatic Cholangiocarcinoma; Extrahepatic Cholangiocarcinoma; Gallbladder Carcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms | interventions — irinotecan sucrosofate; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Irinotecan Liposome Injection + 5-FU/LV (Experimental): The patients in cohort 1 will receive irinotecan liposome injection combined with 5-Fluorouracil (5-FU) and Leucovorin (LV) intravenously on days 1 of every 14-day cycle until disease progression or unacceptable toxicity, or termination of the study for other reasons.
  Interventions: Drug: Irinotecan Liposome Injection; Drug: Fluorouracil; Drug: Leucovorin
- Cohort 2: Irinotecan Liposome Injection + SG001 + 5-Fu/LV (Experimental): The patients in cohort 1 will receive irinotecan liposome injection combined with SG001, 5-Fluorouracil (5-FU) and Leucovorin (LV) intravenously on days 1 of every 14-day cycle until disease progression or unacceptable toxicity, or until 24 months is reached, or the study is terminated for other reasons.
  Interventions: Drug: Irinotecan Liposome Injection; Drug: SG001; Drug: Fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: Irinotecan Liposome Injection — Irinotecan Liposome Injection, intravenously, over 90 min on days 1 of every 14-day cycle, 43mg/10mL
Drug: SG001 — Recombinant Anti-PD-1 Fully Human Monoclonal Antibody Injection, intravenously, over 60 min on days 1 of every 14-day cycle, 100mg/10mL
  Arms: Cohort 2: Irinotecan Liposome Injection + SG001 + 5-Fu/LV
Drug: Fluorouracil — 5-Fluorouracil (5-Fu), intravenously, over 46 h on days 1 of every 14-day cycle
Drug: Leucovorin — Leucovorin (LV), intravenously, over 30 min on days 1 of every 14-day cycle

SUMMARY:
This study is an open-label, phase II study of irinotecan liposome injection in patients with advanced biliary tract cancer. The purpose of this study is to evaluate the safety, efficacy and pharmacokinetics of irinotecan liposome injection in patients with advanced biliary tract cancer.

DETAILED DESCRIPTION:
This is an open-label, parallel, multicentre, phase II study to evaluate the efficacy and safety of irinotecan liposome injection. Eligible patients will be divided into two cohorts according to the criteria for the corresponding cohort. The patients in cohort 1 will receive irinotecan liposome injection combined with 5-Fluorouracil (5-FU) and Leucovorin (LV). The patients in cohort 2 will receive irinotecan liposome injection combined with a PD-1 inhibitor, 5-Fluorouracil and Leucovorin.

ELIGIBILITY:
Inclusion Criteria:

* 1. At least 18 years of age, regardless of gender. 2.Histologically or cytologically confirmed unresectable, locally advanced, or metastatic adenocarcinoma of biliary tract, including intrahepatic cholangiocarcinoma (IHCC), extrahepatic cholangiocarcinoma (EHCC) and gallbladder carcinoma (GBC).

  3.At least one measurable lesion according to RECIST 1.1. 4.Previous first-line standard system chemotherapy failed. First-line standard chemotherapy is defined as gemcitabine combined with capecitabine or platinum.

  5.Patients with prior local treatment (embolization, chemoembolization, radiofrequency ablation, or radical radiotherapy) must be completed at least 4 weeks before the first administration of the study drug, palliative decompensated radiotherapy (such as bone metastases) must be completed at least 2 weeks before the first administration of the study drug.

  6.Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1. 7.Life expectancy >3 months. 8.Adverse reactions must recover to grade 1 or baseline according to CTCAE 5.0 (except for toxicity such as alopecia, grade 2 or less sensory neuropathy, etc., which have been judged no safety risk by investigators).

  9.Patients should not receive cell growth factors or blood and platelet transfusion within 7 days before the initiate administration of study drug, and laboratory test should meet the following criteria: neutrophile count ≥1.5×10^9/L;platelet count ≥90×10^9/L; hemoglobin ≥90 g/L or ≥5.6 mmol/L;serum creatinine ≤1.5×ULN or creatinine clearance rate must be ≥ 50 mL/min when serum creatinine >1.0×ULN;total bilirubin ≤1.5×ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN or ≤2.5×ULN if intrahepatic lesions exist;Albumin ≥3 g/dL.

  10. Activated Partial Thromboplastin Time (APTT), International Normalized Ratio (INR) and prothrombin time (PT) ≤1.5 × ULN for patients not receiving therapeutic anticoagulation.

  11.Patients with biliary obstruction or no evidence of persistent infection should receive adequate biliary drainage; active or suspected infections are not allowed.

  12. Female patients with reproductive potential must agree to use adequate contraception from the signing of informed consent to at least 6 months after the study completion and have a negative serum pregnancy test within 7 days before enrollment, and must be non-lactating. Male patients must agree to use medically approved contraception during the study and for 6 months after the study period.

  13. Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* 1. Patients with definite positive NTRK fusion gene. 2. Patients who have received any investigational drug within 4 weeks prior to the first dose of irinotecan liposomes injection.

  3. Patients with definite metastatic encephalopathy. 4. Patients who have received liver transplantation or liver metastases accounted for 50% or more of the total liver volume.

  5. Patients with hepatic encephalopathy. 6. Uncontrolled third lacunar effusion other than ascites (e.g., large pleural or pericardial effusion).

  7. Previous malignancies in the past five years (except radically resected and non-recurring basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder carcinoma, local prostate carcinoma, carcinoma in situ of cervical, or other carcinoma in situ).

  8. History of serious cardiovascular disease. 9. Patients with uncontrolled active bleeding. 10. Gastrointestinal diseases of clinical significance, such as bleeding, inflammation, obstruction, >grade 1 diarrhea, etc.

  11. Patients with definite Gilbert syndrome. 12. Patients who have concomitant use of strong CYP3A4 inducers within 2 weeks prior to the first dose, or strong CYP3A4 inhibitors or strong UGT1A1 inhibitors within 1 week prior to the first dose.

  13. Patients who received systemic glucocorticoids or other immunosuppressive agents within 14 days before the first dose of the study drug.

  14. Patients who have undergone major organ surgery within 4 weeks prior to the first dose of the study drug.

  15. Patients who are hypersensitivity to any component of irinotecan liposome injection or other liposome products.

  16. Patients who are allergic to gemcitabine, cisplatin, fluorouracil or leucovorin or its components.

Additional exclusion criteria for cohort 2:

1. Patients who have received any other antibodies or drugs that act on T-cell synergetic stimulation or checkpoint pathways (including PD-1, PD-L1, CTLA-4 inhibitors, etc.).
2. Patients with a history of severe allergic reactions to monoclonal antibodies and uncontrolled allergic asthma.
3. Patients with active autoimmune disease or a history of autoimmune diseases.
4. History of primary immunodeficiency.
5. Patients who occurred immune related adverse events.
6. History of allogeneic organ or hematopoietic stem cell transplantation.
7. Received live attenuated vaccine within 14 days before screening period or planned to received it during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to six months after the last patient's first administration
  The percentage of patients who achieve a complete response (CR) or partial response (PR) based on the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to six months after the last patient's first administration
  Time from date of the first dose to date of recorded disease progression or death, whichever occurs first
Overall survival (OS) | Up to six months after the last patient's first administration
  Time from date of the first dose to date of death from any cause
Disease Control Rate (DCR) | Up to six months after the last patient's first administration
  The percentage of patients who achieve a CR, PR or stable disease (SD) based on the RECIST 1.1
Duration of Response (DOR) | Up to six months after the last patient's first administration
  Time from first documented response (CR or PR whichever occurs first, based on investigator's assessment per RECIST 1.1) to date of disease progression or death due to any cause, whichever occurs first
Incidence of treatment-related adverse events (AEs) and serious adverse events (SAEs) | Up to six months after the last patient's first administration
  The AEs and SAEs will be assessed according to the National Cancer Institute (NCI) CTCAE v5.0
Peak Plasma Concentration | 0-240 h of circle 1 to circle 4
  Cmax
Area under the plasma concentration versus time curve | 0-240 h of circle 1 to circle 4
  AUC
UGT1A1 | Within 3 days before the first dose
  UGT1A1 gene polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Cheng, Principal Investigator — Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital)
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No